CLINICAL TRIAL: NCT03909360
Title: Role of Abdominal Drainage for Laparoscopic Cholecystectomy a Prospective Randomised Study
Brief Title: Drainage or Not for Laparoscopic Cholecystetomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: zyeyLCdrainage
Record Dates: First submitted 2019-03-17; First posted 2019-04-10 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Cholecystitis; Cholecystolithiasis; Polyps Gallbladder; Adenomyosis of Gallbladder
MeSH Terms: conditions — Cholecystitis; Cholecystolithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drainage (Experimental): Placement of subhepatic drainage tube for laparoscopic cholecytetomy
  Interventions: Procedure: drainage tube
- no drainage (No Intervention): no placement of subhepatic drainage tube for laparoscopic cholecytetomy

INTERVENTIONS:
Procedure: drainage tube — sub-hepatic drainage tube for laparoscopic cholecystectomy
  Arms: drainage

SUMMARY:
Surgeons usually choosing drainage tube for laparoscopic cholecystectomy according to their experiences but not guidelines. The investigators design a RCT to evaluate the role of drainage in LC surgery and compare the clinical results between drainage and no drainage.

DETAILED DESCRIPTION:
The investigators design a RCT to evaluate the role of drainage in LC surgery and compare the clinical results between drainage and no drainage.

Compare complications as below betwwen drainage and no drainage groups.

1. VAS
2. Nause and vomiting
3. infection
4. bleeding
5. bile leakage
6. puncture drainage
7. readmission
8. reoperation
9. hospital stay
10. hospital expense

ELIGIBILITY:
Inclusion Criteria:

* age:18-75 years old
* indicated and planed to receive laparoscopic cholecystectomy

Exclusion Criteria:

* cirrohosis Child Grading B and C
* upper abdominal surgery history
* adjustment of surgical name intraoperative

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
bleeding Bile leakage | day 1 to one month post LC operation
  the morbidity of bleeding
  the morbidity of bile leakage
bile leakage | day 1 to one month post LC operation
  the morbidity of bile leakage
Puncture drainage Puncture drainage | day 1 to one month post LC operation
  the percentage of puncture drainage
  Puncture drainage
  Puncture drainage
reoperation Reoperation | day 1 to one month post LC operation
  the percentage of reoperation
readmission | day 1 to one month post LC operation
  the percentage of readmission

SECONDARY OUTCOMES:
hospital stay | day 1 to discharge post LC operation
  hospital stay
Hospitalization expenses | day 1 to discharge post LC operation
  Hospitalization expenses
VAS score | day 1 to discharge post LC operation
  VAS score
Nausea and vomiting | day 1 to discharge post LC operation
  the morbidity of Nausea and vomiting
infection | day 1 to discharge post LC operation
  the morbidity of infection (abdominal, incision,pulmonary,et al)

CONTACTS AND LOCATIONS:
Overall Officials: Jiangtao Li, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu H, Liu D, Zhou D, Wu J, Yu Y, Jin Y, Ye D, Ding C, Zhang X, Huang B, Peng S, Li J. Effectiveness of no drainage after elective day-case laparoscopic cholecystectomy, even with intraoperative gallbladder perforation: a randomized controlled trial. Langenbecks Arch Surg. 2023 Mar 1;408(1):112. doi: 10.1007/s00423-023-02846-z. PMID 36856748